CLINICAL TRIAL: NCT02477566
Title: Comparative Study of Long-acting and Short Acting Triptorelin on Pituitary Down-regulation in Long Protocol in PCOS Patients Who Underwent IVF/ICSI Treatment
Brief Title: Comparative Study of Long-acting and Short Acting Triptorelin in PCOS Patients Who Underwent IVF/ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Reproductive Medicine Center, Drum Tower Hospital Affiliated to Nanjing University Medical College, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BL2014003
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: In Vitro Fertilization; Polycystic Ovary Syndrome
Keywords: pcos; Long acting Triptorelin; Short acting Triptorelin; In Vitro Fertilization
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Long-acting Triptorelin (Experimental): Pituitary down-regulation with Long-acting Triptorelin 1.875mg during the luteal
  Interventions: Drug: Long-acting Triptorelin
- Short-acting Triptorelin (Active Comparator): Pituitary down-regulation with Short-acting Triptorelin 0.1mg/d,x10d, then 0.05mg/d until E2<40pg/ml in serum, was initiated during the luteal phase
  Interventions: Drug: Short-acting Triptorelin

INTERVENTIONS:
Drug: Long-acting Triptorelin — Pituitary down-regulation with Long-acting Triptorelin 1.875mg during the luteal phase
  Other Names: Long-acting Triptorelin on pituitary down-regulation
  Arms: Long-acting Triptorelin
Drug: Short-acting Triptorelin — Pituitary down-regulation with Short-acting Triptorelin 0.1mg/d,x10d, then 0.05mg/d until E2<40pg/ml in serum, was initiated during the luteal phase
  Other Names: Short-acting Triptorelin on pituitary down-regulation
  Arms: Short-acting Triptorelin

SUMMARY:
To test whether long-acting Triptorelin on pituitary down-regulation can improve the clinical pregnancy rate and reduces the incidence of ovarian hyperstimulation syndrome (OHSS) in infertile high-risk patients with polycystic ovaries (PCOs) who underwent in vitro fertilization (IVF) or Intracytoplasmic sperm injection

DETAILED DESCRIPTION:
All patients received standard ovarian stimulation with rFSH under pituitary suppression with GnRH agonist according to a protocol used routinely. The long-acting Triptorelin group use long-acting Triptorelin 1.875mg during the luteal phase on Pituitary down-regulation , the Short acting Triptorelin use short-acting Triptorelin 0.1mg/d,x10d, then 0.05mg/d until E2<40pg/ml in serum, was initiated during the luteal phase. Gonadotrophin stimulation of the ovaries was started when serum E2 concentrations declined to < 40 pg/ml and a vaginal ultrasonographic scan showed an absence of follicles > 10mm diameter. Ovarian stimulation was started wih 150-250 IU/day of recombinant FSH (Gonal F, Serono, Switzerland); the initial dose was determined by clinical judgement of the clinician according to the patients's age, body mass index, basal FSH and E2. Transvaginal ultrasound and E2 measurement were used to monitor follicular growth, and gonadotropin dosages were adjusted accordingly. Ovulation was triggered by intramuscular administration of 5000-10,000 IU of human chorionic gonadotropin (HCG, Ferring Pharmaceuticals) when at least two follicles reached a diameter of 18 mm. Serum HCG value were measured at 12 h after HCG trigger using the immunoassay. Oocytes were retrieved 36 h after the injection of HCG.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients diagnosis by Rotterdam Consensus on Diagnostic Criteria who underwent IVF/ICSI treatment

Exclusion Criteria:

* Patients with poor ovarian reserve,
* immunological disease,
* endometriosis,
* uterine abnormality,
* endometrium thickness < 8mm before embryo transfer,
* fewer than two good-quality embryos available for transfer or patients with inadequate data for analysis were excluded.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2 years
  compare the cinical pregnancy rate between long-acting and short-acting Triptorelin on pituitary down-regulation in PCOS patients who underwent IVF/ICSI treatment

SECONDARY OUTCOMES:
moderate/severe OHSS rate | 2 years
  compare the moderate/severe OHSS rate between long-acting and short-acting Triptorelin on pituitary down-regulation in PCOS patients who underwent IVF/ICSI treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Research Room of Reproductive Medicine, The Outpatient Building of Drum Tower Hospital, Nanjing, Jiangsu, China